CLINICAL TRIAL: NCT02425540
Title: Characterization of Ovarian Masses Unable to Classify With Gynecological Ultrasonography: Value of Pelvic MRI With Perfusion- and Diffusion-weighted Imaging
Acronym: IOTAMRI
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S55783
Record Dates: First submitted 2013-08-14; First posted 2015-04-24 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Undetermined Ovarian Mass
Keywords: Pelvic MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with unclassified ovarian mass
  Interventions: Device: Pelvic MRI

INTERVENTIONS:
Device: Pelvic MRI

SUMMARY:
The aim of the study is to prospectively evaluate the value of pelvic MRI including diffusion- and perfusion-weighted sequences in the selected group of patients that have an undetermined ovarian mass at ultrasound.

ELIGIBILITY:
Inclusion Criteria:

*Any woman with an adnexal mass undetermined by gynecological ultrasound

Exclusion Criteria:

* Any lesion with definite diagnosis by gynecological ultrasound
* Denial or withdrawal of oral informed consent.
* Contra-indication for MRI

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ovarian mass not able to classify by gynecological ultrasound
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of MRI findings with histopathology or 2-years follow-up | 03/2015 to 03/2017 (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals UZ Leuven, Gasthuisberg, Leuven, Vlaams-Brabant, Belgium